CLINICAL TRIAL: NCT05078944
Title: Randomized, Blinded, Sham-Controlled Trial of Acupuncture on the Progression of Mild Alzheimer's Disease
Brief Title: Progress of Mild Alzheimer's Disease in Participants on Acupuncture Versus Sham Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Institute of Acupuncture, Moxibustion and Meridian (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ShanghaiIAMM2021052
Record Dates: First submitted 2021-09-23; First posted 2021-10-15 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease 1
Keywords: Alzheimer's Disease; Electroacupuncture
MeSH Terms: conditions — Alzheimer disease type 1; Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active acupuncture + Donepezil (Experimental): Active acupuncture treatment is to be taken 3 sessions weekly over a period of 14 weeks. Donepezil hydrochloride (5 mg/capsule, Weicai Pharmaceutical Co., Ltd, China) is to be taken 5 mg daily over 32 weeks (including 4-week run-in) Intervention: Device: Acupuncture + Drug: Donepezil hydrochloride
  Interventions: Device: Active acupuncture; Drug: Donepezil Hydrochloride
- Sham acupuncture + Donepezil (Sham Comparator): Sham acupuncture treatment with no skin penetration and no current output on sham acupoints is to be taken 3 sessions weekly over a period of 14 weeks. Donepezil hydrochloride (5 mg/capsule, Weicai Pharmaceutical Co., Ltd, China) is to be taken 5 mg daily over 32 weeks (including 4-week run-in) Intervention: Device: Sham acupuncture + Drug: Donepezil hydrochloride
  Interventions: Device: Sham acupuncture; Drug: Donepezil Hydrochloride

INTERVENTIONS:
Device: Active acupuncture — Acupoints: Principal: GV20, EX-HN1, GV24 and bilateral PC6, HT7, ST36, KI3, SP6. Additional: CV6 and bilateral GB39, ST40, SP10 Sterile stainless steel disposable acupuncture needles (size 0.30 × 50 mm, Hwato brand, China) are used. After sterilization, a small plastic ring will be fixed over the acupuncture point with plaster to facilitate maintenance of blinding for the participant, and then the needle will be inserted through the plaster inside the ring. The electric stimulator (SDZ-Ⅲ electroacupuncture apparatus, Hwato brand, China) is applied to GV20, GV24, bilateral PC6 and HT7, dilatational wave, 10/50 Hz and tolerable electric current. Needles placed in other acupoints will be manually stimulated by rotation every 15 minutes. Each session lasts for 45 min.
  Arms: Active acupuncture + Donepezil
Device: Sham acupuncture — Sham acupoints: SA1 (5 cun lateral to GV5), SA2 (5 cun lateral to GV4), SA3 (1 cun lateral to BL56).
  After sterilization, pragmatic placebo needles with blunt tip (size 0.30 × 50 mm, Hwato brand, China) are used. When their tips are pressed against the skin through plastic rings, participants will feel a pricking sensation. The electric stimulator is applied to bilateral SA1 and SA2 with no current output. The mental wire has been cut off with a same outlook as the electroacupuncture group. Needles placed in SA3 will be manually rotated every 15 minutes. Each session lasts for 45 min.
  Arms: Sham acupuncture + Donepezil
Drug: Donepezil Hydrochloride — Donepezil hydrochloride (5 mg/capsule, Weicai Pharmaceutical Co., Ltd, China) is to be taken 5 mg daily.

SUMMARY:
To determine if adjunctive acupuncture acts as an AD treatment rather than a placebo.

DETAILED DESCRIPTION:
Acupuncture is used as an adjuvant therapy for Alzheimer's disease (AD), but available evidence for efficacy is weak. The aim is to determine if adjunctive acupuncture acts as an AD treatment rather than a placebo.

This is a randomized, participant-masked, sham-controlled trial. One hundred and sixty participants with mild AD will be randomly assigned (1:1) to either active acupuncture or non-penetrating sham acupuncture (3 times weekly for 14 weeks) added to donepezil treatment (5 mg per day for 28 weeks). The primary efficacy outcome is the change from baseline in the Alzheimer's disease Assessment Scale (ADAS-cog12). Secondary efficacy outcomes include other assessments of the Mini-Mental State Examination (MMSE), the Alzheimer's disease Cooperative Study-Activities of Daily Living (ADCS-ADL), Neuropsychiatric Inventory (NPI).

ELIGIBILITY:
Inclusion Criteria:

* Meets the diagnostic criteria for probable AD according to the National Institute of Neurological and Communicative Disorders and Stroke/Alzheimer's Disease and Related Disorders Association (NINCDS/ADRDA)
* Scored 1.0 by the Clinical Dementia Rating Scale (CDR) Global Score

Exclusion Criteria:

* Dementia due to other causes
* Evidence of a clinically relevant or unstable psychiatric disorder
* Has irritable bowel syndrome or inflammatory bowel disease
* Has unstable or severe cardiovascular, hepatic, renal, respiratory, endocrinologic, neurologic diseases and other conditions that, in the investigator's opinion, could interfere with the analyses of safety and efficacy in this study
* Has visual or hearing disorder, defeating completion of evaluation
* Use of AD therapy (except for donepezil hydrochloride) which cannot be stopped
* Use of antibiotics within 1 month prior to enrollment
* Has a history of gastrointestinal surgery (except for appendicitis and hernia surgery)
* Without a reliable caregiver who will accompany the participant during treatment and assessment, and monitor administration of the prescribed medications
* With cardiac pacemaker or metal allergy
* Once experienced electroacupuncture treatment before at any time (manual acupuncture is allowed)
* Premenopausal woman

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-06-30 (Actual); Primary Completion 2025-09-10 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Alzheimer's Disease Assessment Scale-Cognitive 12 Item Subscore (ADAS-Cog12) | Baseline, Week 7, Week 14, Week 21, Week 28
  The ADAS is a rater administered instrument that was designed to assess the severity of the dysfunction in the cognitive and noncognitive behaviors characteristic of persons with AD. The cognitive subscale of the ADAS consists of 12 items (ranges from 0 to 75). Higher scores indicating greater cognitive impairment.

SECONDARY OUTCOMES:
Change From Baseline in Mini-Mental State Examination (MMSE) | Baseline, Week 7, Week 14, Week 21, Week 28
  MMSE is a brief screening instrument used to assess cognitive function (orientation, memory, attention, ability to name objects, follow verbal/written commands, write a sentence, and copy figures) in elderly participants. Total score ranges from 0 to 30; lower score indicates greater disease severity.
Change From Baseline in Alzheimer's Disease Cooperative Study Activities of Daily Living (ADCS-ADL) | Baseline, Week 7, Week 14, Week 21, Week 28
  The ADCS-ADL is a 23-item inventory developed as a rater-administered questionnaire answered by the participant's caregiver. The ADCS-ADL measures both basic and instrumental activities of daily living by participants. The total score ranges from 0 to 78, with lower scores indicating greater disease severity.
Change From Baseline in Neuropsychiatric Inventory (NPI) | Baseline, Week 7, Week 14, Week 21, Week 28
  NPI assesses psychopathology in participants with dementia and other neurologic disorders. Information is obtained from a caregiver familiar with the participant's behavior. Total score ranges from 0 to 144, with lower scores indicating fewer behavioral disturbances
Treatment credibility | Week 1, Week 14
  The treatment credibility scale will be assessed by asking participants to rate their response to four questions on a 5-point scale developed by Borkovec and Nau. Total score ranges from 0 to 20; higher score indicates greater treatment credibility.
Incidence of adverse events | Week -4 to Week 28
  Including subcutaneous hematoma, local errhysis at acupoints, sharp pain, palpitation, nausea, dizziness and faint during acupuncture.
Change in gut microbiota diversity based on 16S rRNA gene sequencing analysis | Baseline, Week 14, Week 28
  Stool samples will be processed to extract DNA, followed by 16S rRNA gene sequencing analysis using QIIME and R packages (v3.2.0).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaopeng Ma, MD, PhD, Study Chair — Shanghai Institute of Acupuncture, Moxibustion and Meridian
Locations (1):
- Shanghai Institute of Acupuncture, Moxibustion and Meridian Organization, Shanghai, China

REFERENCES:
- [Derived] Kong X, Ma Z, Tang R, Wang X, Wei K, Yang G, Yang Y, Zhao Y, Zhang D, Xie C, Wang G, Ma X. Efficacy of acupuncture in patients with mild Alzheimer's disease and its impact on gut microbiota: Study protocol for a randomized sham-controlled trial. Front Med (Lausanne). 2023 Feb 23;10:1014113. doi: 10.3389/fmed.2023.1014113. eCollection 2023. PMID 36910501